CLINICAL TRIAL: NCT00937534
Title: An Open Label, Single-dosing, and Parallel Study in Healthy Elderly and Young Male Volunteers.
Brief Title: Study to Compare and Assess the Safety and Pharmacokinetic Characteristics After Oral Administration of Fimasartan (BR-A-657∙K) in Healthy Elderly and Young Male Volunteers
Acronym: Fimasartan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Kyungpook National University Hospital (Other); Seoul National University Hospital (Other)
Responsible Party: Choi, Director, Boryung Pharm Co., Inc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A657-BR-CT-104
Record Dates: First submitted 2009-07-06; First posted 2009-07-13 (Estimated); Last update posted 2009-11-04 (Estimated); Status verified 2009-11

CONDITIONS: Essential Hypertension
Keywords: Fimasartan; healthy elderly and young male volunteer; pharmacokinetic
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Active Comparator): Young male healthy volunteer
  Interventions: Drug: Fimasartan
- Part B (Active Comparator): Elderly male healthy volunteer
  Interventions: Drug: Fimasartan

INTERVENTIONS:
Drug: Fimasartan — Fimasartan 240mg/day

SUMMARY:
The purpose of this study is to compare and assess the safety and pharmacokinetic characteristics after oral administration of fimasartan (BR-A-657∙K) in healthy elderly and young male volunteers.

DETAILED DESCRIPTION:
Fimasartan (BR-A-657-K), a selective blocker of AT1 receptor subtype, showed the rapid and potent antihypertensive effect in many hypertensive models.

Phase I study, Fimasartan (BR-A-657-K) 20 mg ~ 480 mg single dosing with healthy subjects, demonstrated that the Fimasartan (BR-A-657-K) was very safe and well tolerated. Another phase I study, Fimasartan (BR-A-657-K) 120mg and 360mg dosing for 7 days, also showed that Fimasartan (BR-A-657-K) was safe and tolerable though one temporal adverse event was observed in high dose.

A open-labeled, single-dosing, parallel Clinical Study to Evaluate pharmacokinetic characteristics after oral administration of fimasartan in healthy elderly and young male volunteers.

22 male healthy volunteers were enrolled during 2 months.

In part A, 240 mg of fimasartan per day was taken once by younger male healthy volunteers in day 1. Then blood and urine samples were collected 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours after administration.

In part B, 240 mg of hydrochlorothiazide per day was taken once by elderly male healthy volunteers in day 1. Then blood and urine samples were collected 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours after administration.

ELIGIBILITY:
Inclusion Criteria:

* age

  * young: 19-45 years
  * elderly: more than 65 years
* sex: male
* body weight: greater than 55 kg

Exclusion Criteria:

* patients with contraindication to angiotensin II receptor antagonist.
* patients with a history of liver, renal, gastrointestinal, hematological or cardiac diseases
* patients with history or diseases which might affect absorption of the drug
* patients with HIV, type B or C hepatitis
* smokers of 20 or more cigarettes per day

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Cmax, AUClast, tmax, t1/2 | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 h